CLINICAL TRIAL: NCT02589639
Title: A 52-week Randomised, Double-blind, Placebo-controlled, Parallel-group, Efficacy and Safety Study of Empagliflozin Once Daily, as an add-on to Insulin in Japanese Patients With Type 2 Diabetes Mellitus With Insufficient Glycaemic Control
Brief Title: Efficacy and Safety Study of Empagliflozin as add-on to Insulin in Japanese Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1245.107
Record Dates: First submitted 2015-10-27; First posted 2015-10-28 (Estimated); Results first posted 2019-03-27 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2018-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin

ARMS (3):
- empagliflozin 10 mg (Experimental)
  Interventions: Drug: Empagliflozin; Drug: Placebo
- empagliflozin 25 mg (Experimental)
  Interventions: Drug: Empagliflozin; Drug: Placebo
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Empagliflozin
  Arms: empagliflozin 10 mg; empagliflozin 25 mg
Drug: Placebo
  Arms: placebo
Drug: Placebo — For blinding purposes

SUMMARY:
This is a multi-center, randomised, double-blind, placebo-controlled, parallel-group, efficacy and safety study of empagliflozin as add-on to insulin in Japanese patients with Type 2 Diabetes Mellitus with insufficient glycaemic control

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of type 2 diabetes mellitus
* Patients on diet and exercise regimen who are pre-treated with any insulin therapy alone or in combination with 1 oral antidiabetic drug for at least 12 weeks prior to screening
* Fasting C-peptide must be > 0.5 ng/mL
* HbA1c at screening in Patients who are treated with insulin alone must be >=7.5% and <=10.0%
* HbA1c in Patients who are treated with insulin with 1 oral antidiabetic drug (OAD) must be >=7.0% and <=9.5% at screening, and >=7.5% and <=10.0% at placebo run-in period
* Age at informed consent must be >=20 and <75 years
* BMI at screening must be >22 and <=40 kg/m2
* Further inclusion criteria apply

Exclusion criteria:

* Patients who experience uncontrolled hyperglycaemia before randomization
* Patients who are treated with sulfonylurea whose dose is more than a half of daily maximum approval dose, glucagon-like peptide-1 (GLP-1) analogue, thiazolidinedione and sodium-glucose co-transporter 2 (SGLT-2) inhibitor
* Patients with recent cardiovascular and/or stroke events
* Patients with hepatic and/or renal dysfunction
* Patients who received anti-obesity drugs or other treatment leading to unstable body weight
* Patients who have known allergy or hypersensitivity to insulin and/or empagliflozin
* Pre-menopausal women who are nursing or pregnant
* Further exclusion criteria apply

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2015-10-28 (Actual); Primary Completion 2017-04-18 (Actual); Study Completion 2018-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (48):
- Japan (48):
  - Nakayama Clinic, Aichi
  - Kashiwa City Hospital, Chiba, Kashiwa
  - Kunisaki Makoto Clinic, Fukuoka
  - Saiseikai Fukuoka General Hospital, Fukuoka, Fukuoka
  - Seiwakai Medical Corporation Nagata Hospital, Fukuoka, Yanagawa
  - Saiseikai Maebashi Hospital, Gunma, Maebashi
  - Nippon Kokan Fukuyama Hospital, Hiroshima, Fukuyama
  - Jiyugaoka Yokoyama Naika Clinic, Hokkaido, Obihiro
  - Jiyugaoka Yamada Clinic, Hokkaido, Obihiro
  - Souen Diabetes Clinic, Hokkaido, Sapporo
  - Kotani Diabetes Clinic, Hyogo, Kobe
  - Nishinomiya Municipal Central Hospital, Hyogo, Nishinomiya
  - Noritake Clinic, Ibaraki, Ushiku
  - Yokoi Medical Clinic, Kagawa, I.M., Kagawa
  - Fukumoto clinic, Kagoshima
  - Izuro Imamura Hospital, Kagoshima, Kagoshima
  - Wakamatsu Memorial Hospital, Kagoshima, Satsumasendai
  - STOP DM SUZUKI DIABETES CLINIC, Kanagawa, I.M., Kanagawa, Atsugi
  - Takai Naika Clinic, Kanagawa, Kamakura
  - Kokan Clinic, Kanagawa, Kawasaki
  - Yoshimasa Diabetes & Endocrine Clinic, Kyoto, Kyoto
  - Medical Corporation KEISEIKAI Kajiyama clinic, Kyoto, Kyoto
  - Saka General Clinic, Miyagi, Tagajo
  - North Alps Medical Center Azumi Hospital, Nagano, Kitaazumi-gun
  - Asama Nanroku Komoro Medical center, Nagano, Komoro
  - Abe Clinic, Oita, Oita
  - Tsuyama Chuo Hospital, Okayama, Tsuyama
  - AMC Nishi-umeda Clinic, Osaka
  - Shiraiwa Medical Clinic, Osaka
  - Medical Corporation Kyojinkai Clinic Komatsu, Osaka, Neyagawa
  - Minamiosaka Hospital, Osaka, Osaka
  - OCROM Clinic, Osaka, Suita
  - Ageo Central General Hospital, Saitama, Ageo
  - Medical Corporation Kaishinkai Masunaga Clinic, Saitama, Fujimi
  - Medical Corporation Fusa Shimizu Clinic Fusa, Saitama, Saitama
  - Seiwa Clinic, Tokyo, Adachi-ku
  - Juntendo University Hospital, Tokyo, Bunkyo-ku
  - Chiyoda Houjin Clinic, Tokyo, Chiyoda-ku
  - HDC Atlas Clinic, Tokyo, Chiyoda-ku
  - Fukuwa Clinic, Tokyo, Chuo-ku
  - Tokyo-Eki Center-building Clinic, Tokyo, Chuo-ku
  - Tokyo Center Clinic, Tokyo, Chuo-ku
  - Shin Clinic, Tokyo, Ota-ku
  - Shinjuku Research Park Clinic, Tokyo, Shinjuku-ku
  - Sumida Chuou Hospital, Tokyo, Sumida-ku
  - Sagae City Hospital, Yamagata, Sagae
  - Clinic Sugiyama, Yamagata, Yamagata
  - Yamanashi Prefectural Central Hospital, Yamanashi, Kofu

REFERENCES:
- [Derived] Tuttle KR, Levin A, Nangaku M, Kadowaki T, Agarwal R, Hauske SJ, Elsasser A, Ritter I, Steubl D, Wanner C, Wheeler DC. Safety of Empagliflozin in Patients With Type 2 Diabetes and Chronic Kidney Disease: Pooled Analysis of Placebo-Controlled Clinical Trials. Diabetes Care. 2022 Jun 2;45(6):1445-1452. doi: 10.2337/dc21-2034. PMID 35472672

RESULTS

PARTICIPANT FLOW:
Recruitment Details: After screening, patients who were pre-treated with insulin and 1 oral antidiabetic drug (OAD) underwent a 10-week wash-out period.
  Then patients proceeded to a 2-week open-label placebo run-in period. Patients who were pre-treated with insulin alone skipped the wash-out period and proceeded to an open-label placebo run-in period.
Pre-assignment Details: Patients who successfully completed the periods and who still satisfied the inclusion/exclusion criteria were randomised to the 52-week double- blind treatment period of the study in which they received either 1 of the 2 doses of empagliflozin or placebo in addition to insulin.
Groups:
- Placebo: Patients were orally administered Placebo matching Empagliflozin 10 milligram (mg) or 25 mg once daily for 52 weeks of double-blind treatment period
- Empagliflozin 10 mg: Patients were orally administered Empagliflozin 10 mg film-coated tablet once daily for 52 weeks of double-blind treatment period
- Empagliflozin 25 mg: Patients were orally administered Empagliflozin 25 mg film-coated tablet once daily for 52 weeks of double-blind treatment period
Period: Overall Study
Arm/Group | Placebo | Empagliflozin 10 mg | Empagliflozin 25 mg
Started | 90 | 89 | 90
Treated | 90 | 86 | 90
Completed | 80 | 79 | 86
Not Completed | 10 | 10 | 4
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Patient withdrawal, not due to AE | 3 | 0 | 0
Not completed — Adverse Event | 4 | 5 | 3
Not completed — Other reason than specified above | 1 | 2 | 1
Not completed — Not Treated | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) consisted of all patients in the treated set (TS) who had a baseline measurement of the primary endpoint.
  (The treated set (TS) consisted of all randomised patients who were treated with at least 1 dose of the study drug during the 52-week double blind treatment period. The TS was the basis for safety analyses)
Groups:
- Total: Total of all reporting groups
Arm/Group | Empagliflozin 10 mg | Empagliflozin 25 mg | Placebo | Total
Number analyzed (Participants) | 90 | 86 | 90 | 266
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (10.7) | 58.3 (10.0) | 58.6 (9.5) | 58.7 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 23 | 29 | 73
  Male | 69 | 63 | 61 | 193
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Baseline glycosylated haemoglobin A1c (HbA1c) [%] [Mean (Standard Deviation); unit: % of HbA1c] | 8.70 (0.68) | 8.83 (0.66) | 8.74 (0.72) | 8.75 (0.69)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Haemoglobin A1c (HbA1c) After 16 Weeks of Treatment.
Description: The primary endpoint was the change from baseline in HbA1c after 16 weeks of treatment.
  The term "baseline" refers to the last observation prior to the administration of any randomised study drug.
  Means presented are the adjusted means.
Time Frame: Baseline and 16 weeks
Population: Full analysis set (FAS) with last observation carried forward at 16 weeks (LOCF)-16; The FAS consisted of all patients in the TS who had a baseline measurement of the primary endpoint.
Measure: Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Placebo | Empagliflozin 10 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 90 | 86 | 90
percentage of HbA1c | 0.00 (0.07) | -0.92 (0.07) | -1.00 (0.07)
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 mg; The statistical model was: Change from baseline in HbA1c after 16 weeks = overall mean + baseline HbA1c + treatment + baseline renal function + type of insulin therapies + random error; Test type: Superiority — The superiority of empagliflozin 10 mg against placebo was tested for change from baseline in HbA1c after 16 weeks of treatment at the level of α=0.05 (2-sided); p < 0.0001, ANCOVA; Analysis of Covariance (ANCOVA) comparing the change from baseline in HbA1c after 16 weeks of treatment; Mean Difference (Final Values) = -0.92, 95% CI 2-sided [-1.11 to -0.73], Standard Error of Mean 0.09; Adjusted Mean Difference calculated as (Empagliflozin 10 mg - Placebo)
Statistical Analysis 2: Comparison: Placebo vs Empagliflozin 25 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — The superiority of empagliflozin 25 mg against placebo was tested for change from baseline in HbA1c after 16 weeks of treatment at the level of α=0.05 (2-sided); p < 0.0001, ANCOVA; Analysis of Covariance (ANCOVA) comparing the change from baseline in HbA1c after 16 weeks of treatment; Mean Difference (Final Values) = -1.00, 95% CI 2-sided [-1.18 to -0.82], Standard Error of Mean 0.09 — Adjusted Mean Difference calculated as (Empagliflozin 10 mg - Placebo)

2. Secondary Outcome: Percentage of Patients With Investigator Defined Drug-Related Adverse Events (AEs)
Description: Percentage of patients with investigator defined drug-related Adverse Events (AEs) are presented
Time Frame: From 1st intake of study drug to last intake of study drug + 7 days; up to 53 weeks
Population: Treated set (TS): TS consisted of all randomised patients who were treated with at least 1 dose of the study drug during the 52-week double blind treatment period. The TS was the basis for safety analyses.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Empagliflozin 10 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 90 | 86 | 90
Percentage of participants | 25.6 | 43.0 | 43.3

ADVERSE EVENTS:
Time Frame: From 1st intake of study drug to last intake of study drug + 7 days; up to 53 weeks
Arm/Group | Placebo | Empagliflozin 10 mg | Empagliflozin 25 mg
All-Cause Mortality (participants affected / at risk) | 0/90 | 1/86 | 0/90
Serious Adverse Events (participants affected / at risk) | 6/90 | 9/86 | 8/90
Other Adverse Events (participants affected / at risk) | 49/90 | 45/86 | 48/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=90) | Empagliflozin 10 mg (N=86) | Empagliflozin 25 mg (N=90)
Arthritis bacterial (Infections and infestations) | 0 | 1 | 0
Chronic sinusitis (Infections and infestations) | 0 | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0
Vocal cord paralysis (Nervous system disorders) | 0 | 1 | 0
Glaucoma (Eye disorders) | 0 | 0 | 2
Cataract (Eye disorders) | 0 | 0 | 1
Dyschromatopsia (Eye disorders) | 0 | 0 | 1
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=90) | Empagliflozin 10 mg (N=86) | Empagliflozin 25 mg (N=90)
Nasopharyngitis (Infections and infestations) | 28 | 30 | 24
Asymptomatic bacteriuria (Infections and infestations) | 8 | 3 | 5
Hypoglycaemia (Metabolism and nutrition disorders) | 19 | 24 | 25
Eczema (Skin and subcutaneous tissue disorders) | 5 | 5 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 5 | 6
Pollakiuria (Renal and urinary disorders) | 2 | 9 | 9
Blood ketone body increased (Investigations) | 1 | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2016-09-13): https://cdn.clinicaltrials.gov/large-docs/39/NCT02589639/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-26): https://cdn.clinicaltrials.gov/large-docs/39/NCT02589639/SAP_001.pdf